CLINICAL TRIAL: NCT06940947
Title: Endoscopic THerapy Or Surgery for Early Colon Cancer (ETHOS)
Brief Title: Endoscopic Therapy Or Surgery for Early Colon Cancer
Acronym: ETHOS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Norwegian Department of Health and Social Affairs (Other Government)
Collaborators: Medical University of Gdansk (Other); Vestre Viken Hospital Trust (Other); Medical Biometry and Epidemiology_- Universitätsklinikum Hamburg Eppendorf (Unknown); Institute of Oncology in Warsaw (Unknown); Karolinska Institutet (Other); University Hospital, Limoges (Other); University Hospital, Akershus (Other); University of Roma La Sapienza (Other); Hospital Clinic of Barcelona (Other); Leuven University Medical Center (Unknown); University Hospital, Ghent (Other); Sørlandet Hospital (Unknown); Northern Norway Regional Health Trust (Unknown); Helse Stavanger HF (Other Government); Haukeland University Hospital (Other); St. Olavs Hospital (Other); University of Oslo (Other); Frontier Science Foundation (Unknown)
Responsible Party: Principal Investigator, Michael Bretthauer, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 840389
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eFTR (Experimental): endoscopic full thickness resection
  Interventions: Procedure: eFTR
- Surgery (Active Comparator): standard-of-care surgery
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: eFTR — endoscopic full thickness resection
  Arms: eFTR
Procedure: Surgery — standard-of-care surgery
  Arms: Surgery

SUMMARY:
The trial is a randomized head-to-head comparison of the benefits, harms and burdens of endoscopic full-thickness resection (eFTR), a novel, minimally invasive endoscopic treatment modality, for early colon cancer as compared to standard-of-care surgery.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed biopsy-confirmed colon cancer (adenocarcinoma) with macroscopic suspicion of submucosal invasion considered removable by EFTR as deemed by the local multidisciplinary team (MDT) at the participating center
* Size ≤20 mm in diameter as deemed by the colonoscopist
* No presence of histopathological high-risk features in biopsy (high grade tumor growth, budding grade 2 or 3, or lymphovascular invasion)
* Patient eligible for surgical removal as deemed by the local MDT at the participating center
* Endoscopic images or video of the tumor
* No sign of disease beyond T2N0M0 on pre-treatment imaging, biopsy sampling, and radiographic and clinical evaluation
* No contraindication for any of the two treatment arms
* Written informed consent
* No prior or synchronous CRC
* No other malignancy which is not cured
* No more than 10 adenomas or serrated polyps
* No genetic cancer syndrome (adenomatous or serrated polyposis syndrome; Lynch or Lynch-like syndrome)
* No inflammatory bowel disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 434 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2033-09-01 (Estimated); Study Completion 2033-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of severe adverse events, re-admissions and deaths within 30 days | 30 days
  co-primary short-term endpoint is the composite rate of rate of severe adverse events, re-admissions and deaths within 30 days following assigned treatment
Rate of cancer recurrence or CRC death after three years | 3 years
  primary long-term endpoint of CRC death or cancer recurrence or sign of lymph nodes or distant metastases after three years

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Gdańsk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Yes
Only if ethical approval is granted by the other researchers, and the study scientific board has reviewed and approved the proposal